CLINICAL TRIAL: NCT00954980
Title: Evaluation of Clinical Characteristics of Endovenous Sclerotherapy of Varicose Veins
Brief Title: Evaluation of Endovenous Sclerotherapy for Treatment of Varicose Veins
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Suman Rathbun, Professor of Medicine, University of Oklahoma
Other Study IDs: 14632; 20091634 (Other: Office of Research Administration)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Varicose Veins
Keywords: Varicose Veins; Superficial Thrombophlebitis; Deep Vein Thrombosis; Ulceration; leg pain; leg swelling
MeSH Terms: conditions — Varicose Veins; Venous Thrombosis; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples will be obtained for measurement of D-dimer, fibrin monomer, and total microparticles.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endovenous Sclerotherapy: For those who have been diagnosed with varicose veins of the leg and have been scheduled to undergo an endovenous sclerotherapy procedure

SUMMARY:
The overall objective will be to evaluate clinical predictors of outcomes in patients who undergo endovenous sclerotherapy for the treatment of varicose veins.

DETAILED DESCRIPTION:
A prospective cohort study of patients who undergo endovenous sclerotherapy over 2 years. There are no deviations in usual clinical assessment and care of patients seeking varicose vein treatment. The purpose of this protocol is only to collect clinical and biomarker information related to this standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of varicose veins

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vascular or primary care clinic patients who have been scheduled to undergo an endovenous sclerotherapy procedure
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of obliteratin (total or partial) of injected varicosity. | assessment will be at 1, 12, and 26 weeks.
Improvement in venous stasis symptoms. | assessment will be at 1, 12, and 26 weeks
Change in quality of life. | assessment will be at 1, 12, and 26 weeks
Associations between clinical outcomes and biomarkers. | assessment will be at 1, 12, and 26 weeks

SECONDARY OUTCOMES:
Recurrence of varicosities. | assessment will be at 1, 12, and 26 weeks
Adverse events reported following procedure. | assessment will be at 1, 12, and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suman W. Rathbun, M.D., Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- University of Oklahoma Health Sciences Center campus at the OU Vascular Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided